CLINICAL TRIAL: NCT02774564
Title: Pharmacokinetic-pharmacodynamic Interaction Between Three Different Single Doses of BIA 3-202 and a Single Dose of Controlled-release 200/50 mg Levodopa/Carbidopa (Sinemet® cr 200/50): a Double-blind, Randomised, Four-way Crossover, Placebo-controlled Study in Healthy Volunteers
Brief Title: Pharmacokinetic-pharmacodynamic Interaction Between BIA 3-202 and Levodopa/Carbidopa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-107
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nebicapone 50 mg (Experimental): 1 tablet of 50 mg plus 3 tablets of placebo concomitantly with 1 tablet of Sinemet® CR 200/50 (levodopa 200 mg / carbidopa 50 mg)
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: Sinemet®
- Nebicapone 100 mg (Experimental): 2 tablets of 50 mg plus 2 tablets of placebo concomitantly with 1 tablet of Sinemet® CR 200/50 (levodopa 200 mg / carbidopa 50 mg)
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: Sinemet®
- Nebicapone 200 mg (Experimental): 4 tablets of 50 mg concomitantly with 1 tablet of Sinemet® CR 200/50 (levodopa 200 mg / carbidopa 50 mg)
  Interventions: Drug: BIA 3-202; Drug: Sinemet®
- Placebo (Placebo Comparator): 4 tablets concomitantly with 1 tablet of Sinemet® CR 200/50 (levodopa 200 mg / carbidopa 50 mg)
  Interventions: Drug: Placebo; Drug: Sinemet®

INTERVENTIONS:
Drug: BIA 3-202 — Nebicapone tablets 50 mg, oral administration
  Other Names: Nebicapone
  Arms: Nebicapone 100 mg; Nebicapone 200 mg; Nebicapone 50 mg
Drug: Placebo — Nebicapone matching placebo tablets
  Arms: Nebicapone 100 mg; Nebicapone 50 mg; Placebo
Drug: Sinemet® — Sinemet® CR 200/50 (levodopa 200 mg / carbidopa 50 mg) tablets

SUMMARY:
The purpose of this study is to the effect of three single oral doses of nebicapone (50 mg, 100 mg and 200 mg) on the levodopa pharmacokinetics when administered in combination with a single-dose of controlled release levodopa 200 mg/carbidopa 50 mg (Sinemet CR 200/50).

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled, 4-way crossover study with four single-dose treatment periods. The washout period between doses was 5 days or more.

Procedures:

Screening: Subjects will be screened for eligibility within 28 and 7 days of first admission. Written informed consent will be obtained before any study procedure is performed. The screening will consist of: medical history; physical examination, vital signs; complete neurological examination; 12-lead ECG; hematology, coagulation, plasma biochemistry and urinalysis tests; HIV, hepatitis B and hepatitis C serology; drugs of abuse and alcohol screen; urine pregnancy test in women of childbearing potential; and review of the selection criteria. The results of screening must be known to the investigator prior to the subject's first admission.

Treatment periods: In each of the four consecutive treatment periods, eligible subjects will be admitted to the UFH on the day prior to receiving the study medication for: vital signs; medical history and physical examination updates; 12-lead ECG; hematology and plasma biochemistry; drugs of abuse and alcohol screen; and urine pregnancy test in women of childbearing potential. On the first admission the subjects will have a review of the selection criteria and will be randomized to one of the treatment sequences. On the morning of the dosing day, subjects will receive a dose of BIA 3-202 / Placebo concomitantly with a dose of Sinemet CR 200/50 in fasting conditions (at least 8 hours) and will remain in the UFH until at least 24 h post-dose; then, they will be discharged and will return for the next period or the follow-up visit. At given time-points between pre-dose and discharge, subjects will be submitted to vital signs recording, brief neurological examinations, 12-lead ECG, and blood sampling for plasma drug assays and erythrocyte S-COMT activity. At discharge, vital signs and ECG will be recorded, and hematology and plasma biochemistry tests will be performed.

Follow-up: A follow-up visit will occur approximately 7-10 days after discharge of the last treatment period or early discontinuation for: medical history and physical examination updates; vital signs; 12-lead ECG; hematology, plasma biochemistry and urinalysis tests; and pregnancy test in women of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for entry into the study if they fulfilled the following inclusion criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission to first treatment period.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Subjects who were non-smokers or who smoked ≤ 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

Subjects were not eligible for entry into the study if they fulfilled the following exclusion criteria:

* Subjects who did not conform to the above inclusion criteria, or
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of glaucoma.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or first admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used medicines within 2 weeks of first admission that, in the opinion of the investigator, may affect the safety or other study assessments.
* Subjects who had used any investigational drug or participated in any clinical trial within 2 months of their first admission.
* Subjects who had donated or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
  Cmax - Maximum observed plasma concentration of levodopa following oral administration of single-doses of Sinemet® CR 200/50 concomitantly with placebo or nebicapone
Tmax | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
  Tmax - Time to occurrence of Cmax of levodopa following oral administration of single-doses of Sinemet® CR 200/50 concomitantly with placebo or nebicapone
AUC0-t | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
  AUC0-t - Area under the plasma concentration-time curve from time 0 to the last sampling time at which concentration were at or above the Limit of quantification of levodopa following oral administration of single-doses of Sinemet® CR 200/50 concomitantly with placebo or nebicapone
AUC0-∞ | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
  AUC0-∞ - Area under the plasma concentration-time curve extrapolated to infinity of levodopa following oral administration of single-doses of Sinemet® CR 200/50 concomitantly with placebo or nebicapone

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit, S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided